CLINICAL TRIAL: NCT01116167
Title: Letrozole and Berberine in Infertile PCOS Patients
Brief Title: Polycystic Ovary Syndrome (PCOS): Effect Of Letrozole and Berberine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heilongjiang University of Chinese Medicine (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Xiaoke Wu, Professor and Department Chairman of Obstetrics and Gynecology, Heilongjiang University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: you070316
Record Dates: First submitted 2010-04-27; First posted 2010-05-04 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Letrozole; Berberine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Letrozole -Berberine (Experimental)
  Interventions: Drug: Letrozole -Berberine
- Letrozole (Active Comparator)
  Interventions: Drug: Letrozole
- Berberine (Active Comparator)
  Interventions: Drug: Berberine

INTERVENTIONS:
Drug: Letrozole -Berberine — Letrozole
  2.5 mg letrozole daily from day 5 of the menses for 5 days for month 1 to 3, 5.0 mg letrozole daily from day 5 of the menses for 5 days for month 4 to 6.
  Berberine
  1.5g daily for 6 month.
  Arms: Letrozole -Berberine
Drug: Letrozole — Letrozole
  2.5 mg letrozole daily from day 5 of the menses for 5 days for month 1 to 3, 5.0 mg letrozole daily from day 5 of the menses for 5 days for month 4 to 6.
  Berberine Placebo
  5 tablet tds for 6 months
  Arms: Letrozole
Drug: Berberine — Berberine
  1.5g daily for 6 month.
  Letrozole placebo
  1 tablet daily from day 5 of the menses for 5 days for month 1 to 3, 2 tablets daily from day 5 of the menses for 5 days for month 4 to 6.
  Arms: Berberine

SUMMARY:
Polycystic ovary syndrome (PCOS) is a heterogeneous disorder affecting almost4%-7% of the female population of reproductive age. Its heterogeneity is characterized by a wide spectrum of features, including ovulatory dysfunction and infertility, hyperandrogenism, hyperinsulinemia, insulin resistance (IR), and progression to type 2 diabetes.Since the Ming Dynasty in China,PCOS has been defined as "phlegm and wetness"infertility in traditional Chinese medicine ,namely "metabolic infertility".Chinese herbs have been used to treat PCOS for thousands of years with good effects.Berberine has also been used for diabetic patients in traditional Chinese medicine for hundreds of years. Recent studies have reported its effects on hyperglycemia and dyslipidemia.The purpose of this study is to determine whether Letrozole combined with berberine are effective in the treatment of infertile PCOS patients.

ELIGIBILITY:
Inclusion Criteria:

* Chinese women
* Age between 20 and 40 years.
* Confirmed diagnosis of PCOS according to the Rotterdam 2003 criteria (2 out of 3):

  1. Oligo- or anovulation
  2. Clinical and/or biochemical signs of hyperandrogenism
  3. Polycystic ovaries and exclusion of other etiologies (congenital adrenal hyperplasia, androgen-secreting tumors, Cushing's syndrome)
* At least one patent tube and normal uterine cavity shown by hysterosalpingogram, HyCoSi or diagnostic laparoscopy within three years.
* Sperm concentration 20×106/mL and progressive motility (grades a and b) ≥50%.

Exclusion Criteria:

* Use of hormonal drugs or other medications including Chinese herbal prescriptions in the past 3 months.
* Patients with known sever organ dysfunction or mental illness.
* Pregnancy, post-abortion or postpartum within the past 6 weeks.
* Breastfeeding within the last 6 months.
* Not willing to give written consent to the study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 660 (Estimated)
Dates: Start 2009-10; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Live-birth rate | Up to 2 years

SECONDARY OUTCOMES:
Ovulation rate | Up to 1 year
Ongoing pregnancy rate at around gestation 8-10 weeks | Up to 1 year
Multiple pregnancy rate | Up to 1 year.
Miscarriage rate: loss of an intrauterine pregnancy before 20 completed weeks of gestation | Up to 1 year
Other pregnancy complications such as early pregnancy loss, gestational diabetes mellitus, pregnancy-induced hypertension and birth of small-for-gestational-age (SGA) babies. | Up to 1 year
Infant outcome | Up to 1 year
Changes in metabolic profile: glucose and insulin concentrations, cholesterol, triglycerides, high density lipoprotein (HDL-C) and low density lipoprotein (LDL-C) | Up to 1 year
Changes in hormonal profile: Follicle-stimulating hormone (FSH), Luteinizing hormone (LH), total testosterone (T), Sex hormone-binding globulin (SHBG) and Dehydroepiandrosterone sulfate (DHEAS) | Up to 1 year
Side effect. | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lihui Hou, MD., Study Chair — The First Affliated Hospital,Heilongjiang University of Chinese Medicine .; Xiaoke Wu, MD.PhD., Study Chair — The First Affliated Hospital,Heilongjiang University of Chinese Medicine
Locations (18):
- China (18):
  - Affiliated Hospital of Anhui University of Chinese Medicine, Hefei, Anhui
  - Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangzhou Medical School First Affiliated Hospital, Guangzhou, Guangdong
  - Daqing LongNa Hospital, Daqing, Heilongjiang
  - Daqing Longnan hospital, Daqing, Heilongjiang
  - Obstetrics and Gynecology,Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang
  - First Affliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Mudanjiang maternal and children hospital, Mudanjiang, Heilongjiang
  - 2nd Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, Henan
  - First Affiliated Hospital of Hunan University of Chinese, Changsha, Hunan
  - SuqianMaternal and Child Health Hospital, Suqian, Jiangsu
  - First Hospital, Jiangxi college of Chinese Medicine, Nanchang, Jiangxi
  - Dalian Maternal and Child Health Hospital, Dalian, Liaoning
  - Shanxi Hospital of Chinese Medicine, Taiyuan, Shanxi
  - First Affiliated Hospital of Tianjin University of Chinese Medicine, Tianjin, Tianjin Municipality
  - Second Affiliated Hospital, Tianjin University of Chinese Medicine, Tianjin, Tianjin Municipality
  - Zhejiang province hospital of integrated traditional and western medicine, Hangzhou, Zhejiang
  - Second Affiliated Hospital of Heilongjiang University of Chinese Medicine, Harbin

REFERENCES:
- [Derived] Zhou K, Zhang J, Xu L, Lim CED. Chinese herbal medicine for subfertile women with polycystic ovarian syndrome. Cochrane Database Syst Rev. 2021 Jun 4;6(6):CD007535. doi: 10.1002/14651858.CD007535.pub4. PMID 34085287
- [Derived] Li Y, Kuang H, Shen W, Ma H, Zhang Y, Stener-Victorin E, Hung E, Ng Y, Liu J, Kuang H, Hou L, Wu X. Letrozole, berberine, or their combination for anovulatory infertility in women with polycystic ovary syndrome: study design of a double-blind randomised controlled trial. BMJ Open. 2013 Nov 25;3(11):e003934. doi: 10.1136/bmjopen-2013-003934. PMID 24282248